CLINICAL TRIAL: NCT03425409
Title: Aviation Portable Oxygen Delivery System Based on Pneumatic Pulse Technology
Brief Title: Aviation Portable Oxygen Delivery System
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Duke University (Other)
Collaborators: Odessey II Solutions (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Device Feasibility
Other Study IDs: Pro00087584
Record Dates: First submitted 2018-01-31; First posted 2018-02-07 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Oxygen Delivery Systems at Altitude

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous Flow (Other): Oxygen delivery at 4 liters per minute is the standard method
  Interventions: Device: Integra Pulse Portable- Continuous flow
- Pneumatic Pulsed Flow (Other): Oxygen delivery using test method
  Interventions: Device: Integra Pulse Portable- Pneumatic pulsed flow

INTERVENTIONS:
Device: Integra Pulse Portable- Continuous flow — 4 liters per minute oxygen flow
  Arms: Continuous Flow
Device: Integra Pulse Portable- Pneumatic pulsed flow — Oxygen flow determined by test device
  Arms: Pneumatic Pulsed Flow

SUMMARY:
This study aims to investigate dose based oxygen delivery vs. continuous flow of oxygen during simulated altitude conditions as would be experienced after a loss of pressure during commercial aircraft flight. Testing will be performed at rest and during light exercise at a simulated altitude of 15,000 feet in a hypobaric chamber. Performance of the two oxygen delivery systems will be compared using oxygen saturation determined by pulse oximetry.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers

Exclusion Criteria:

* smoking
* pregnancy
* sickle cell trait
* cardiovascular or pulmonary disease
* significant ear or sinus problems that would prevent equalization during pressure change
* estimated VO2peak <35 mL/kg per minute (males) or <30 mL/kg per minute (females)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2018-10-01 (Estimated); Study Completion 2018-10-01 (Estimated)

PRIMARY OUTCOMES:
Device performance, as measured by SpO2 | one minute
  The same subject must complete both oxygen delivery system exposures for the data to be used in system performance analysis. Equivalence of the two oxygen delivery systems will be defined as the lack of statistically significant difference (N=20) in SpO2 during the last minute of exercise between the pulse and continuous flow oxygen delivery systems. Average minimum SpO2 over the last minute of the test period will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Moon, MD, Principal Investigator — Duke Universtiy Health System

IPD SHARING:
Plan to Share IPD: No